CLINICAL TRIAL: NCT03102892
Title: Adjuvant Effect of Antimicrobial Photodynamic Therapy on Periodontal Treatment and Salivary Status of Type 1 Diabetes Mellitus Patients
Brief Title: Antimicrobial Photodynamic Therapy on Periodontal Treatment and Salivary Status of Type 1 Diabetes Mellitus Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemics
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Carla Andreotti Damante, Associate professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BauruSchoolDentistryPDTDM1
Record Dates: First submitted 2017-03-30; First posted 2017-04-06 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Diabetes Mellitus, Type 1; Periodontal Diseases; Periodontal Pocket
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Periodontal Diseases; Periodontal Pocket

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scaling Root Planing (Active Comparator): Treatment by scaling and root planing. Repetition after 7 and 14 days.
  Interventions: Procedure: Scaling root planing
- Antimicrobial Photodynamic Therapy (Experimental): Scaling and root planing and Antimicrobial photodynamic therapy with red laser (658 nm, 0.1 Watts, 2229 J/cm², 10s per point) and methylene blue dye (10mg/ml). Repetition after 7 and 14 days.
  Interventions: Procedure: Scaling root planing; Procedure: Antimicrobial photodynamic therapy

INTERVENTIONS:
Procedure: Scaling root planing — Treatment by scaling and root planing alone.
Procedure: Antimicrobial photodynamic therapy — Treatment with methylene blue dye and red laser
  Arms: Antimicrobial Photodynamic Therapy

SUMMARY:
The aim of this study is to evaluate adjuvant effect of antimicrobial photodynamic therapy in periodontal treatment and salivary status of type 1 diabetes patients.

DETAILED DESCRIPTION:
Diabetes Mellitus is a risk factor for periodontal disease increasing its prevalence, extension and severity. Periodontal disease is considered the sixth complication of diabetes. There is a global epidemic of diabetes, including an increase of type 1 diabetes incidence in younger patients. Adjuvant treatments to scaling and root planing as antimicrobial photodynamic therapy show improved clinical outcomes. Thus, the aim of this randomized clinical trial is to evaluate adjuvant effect of antimicrobial photodynamic therapy in periodontal treatment and salivary status of type 1 diabetes patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnose of Type 1 diabetes mellitus
* Age between 18 to 65 years old
* Presence of at least one tooth for hemiarch
* Moderate and severe periodontal disease

Exclusion Criteria:

* Type 2 diabetes mellitus
* Total edentulism
* Smokers
* Pregnancy
* Systemic diseases as other endocrine diseases and blood diseases
* Use of drugs that alter periodontal tissue as phenytoin and cyclosporine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Periodontal disease (gingivitis and periodontitis) measured by a periodontal probe and classified according to severity | 6 months
  Severe periodontitis was defined by the presence of ≥ 2 interproximal sites in different teeth with clinical attachment level (CAL) ≥ 6mm and ≥1 interproximal site with periodontal probing depth (PPD) ≥5mm. Moderate periodontitis was defined by the presence of ≥ 2 interproximal sites in different teeth with CAL ≥ 4mm or ≥ 2 interproximal sites in different teeth with PPD ≥5mm. Mild periodontitis was defined as ≥ 2 interproximal sites in different teeth with ≥ 3 mm CAL and ≥ 2 interproximal sites in different teeth with ≥ 4 mm PPD or at least 1 site with PPD ≥ 5 mm (20,21). Gingivitis was determined as follows: Subjects were considered healthy if presented PPD ≤3mm/Bleeding on probing (BOP) extent scores < 10% and with gingivitis if presented PPD ≤3mm/ BOP extent scores >10%.
Salivary glucose - collection of stimulated saliva in 10 minutes and measured with a colorimetric kit | 6 months
  Salivary glucose is measured by a colorimetric kit and the values are converted and presented as mg/dL. There are no reference value for this measurement. The analysis is done by means of correlation to blood glucose levels in mg/dL.

SECONDARY OUTCOMES:
Salivary pH and buffering Capacity - collection of stimulated saliva in 10 minutes and measurement of acidity with a pHmeter | 6 months
  Normal Salivary pH = 6 to 7. Buffering capacity: ≥ 5.6 were considered as ''high'', ranging from 4.1 to 5.5 were labelled as ''medium'' and those ≤4 were defined as ''low''.
Capillary glycemia measured by a glucometer | 6 months
  Normal glycemia: <100mg/dL

CONTACTS AND LOCATIONS:
Locations (1):
- Bauru School of Dentistry, Bauru, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Zahrani MS, Bamshmous SO, Alhassani AA, Al-Sherbini MM. Short-term effects of photodynamic therapy on periodontal status and glycemic control of patients with diabetes. J Periodontol. 2009 Oct;80(10):1568-73. doi: 10.1902/jop.2009.090206. PMID 19792844